CLINICAL TRIAL: NCT01196533
Title: A Comparative Clinical Trial to Assess the Accuracy of the TensorTip, a Novel Non Invasive Device for the Measurement of Physiological and Blood Chemistry Parameters
Brief Title: A Comparative Clinical Trial of the TensorTip, a Novel Non Invasive Device for Measurement Blood Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cnoga Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CMIL-MHUS-V1.0
Record Dates: First submitted 2010-08-29; First posted 2010-09-08 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-07

CONDITIONS: Anemia; Diabetes; Heart Disease; High Blood Pressure; Hypotension; Metabolic Diseases; Respiratory Diseases
MeSH Terms: conditions — Anemia; Diabetes Mellitus; Heart Diseases; Hypertension; Hypotension; Metabolic Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non Invasive Monitoring (Experimental): Intervention: Device: Non invasive peripheral blood monitoring
  Interventions: Device: Non invasive peripheral blood monitoring

INTERVENTIONS:
Device: Non invasive peripheral blood monitoring — non invasive monitoring

SUMMARY:
1. Aim:

   The aim of the clinical trial is to study the accuracy of the TensorTip device compared with registered (FDA-approved) invasive and non-invasive devices.
2. Hypothesis:

Human physiological biomarkers may be measured from the color distribution of the internal or external (skin) tissue. The technology of the TensorTip finger-mounted device is based on the color distribution of the peripheral blood tissue, which enables the measurement of certain biomarkers and vital signs under consideration.

DETAILED DESCRIPTION:
The TensorTip (previously named Soft Touch) is a novel non invasive Finger tip device that. The Tensor Tip is a non-invasive device which was designed and aimed to measure a wide range of physiological and bio-parameters such as blood glucose, hemoglobin and hematocrit, blood PH, oxygen saturation SpO2, blood carbon dioxide, blood pressure, peripheral pulse and more based on the temporarily color distribution of the tissue under consideration. The Tensor Tip is based on real time color image sensor, real time photographing the fingertip tissue. A color image sensor of the type used in the Tensor Tip enables a wide range of information in the spectral, resolution, dynamic range and time domains enabling further investigation of the blood chromatic changes as a function body physiology. The concept behind this investigation reflects the idea that a change in human physiology condition would temporarily change the blood pigmentation.

The present study is aimed to assess the accuracy of the novel device in measuring all the above mentioned parameters by recording AS IS the change of the fingertip color tissue while simultaneous recording the standard invasive measured parameters on daily or periodic routine in the hospitalized patients.

This vast data recordings (tissue and references) enable the Tensor tip to analyze a particular bio parameter. The tensor tip is calibrated to a certain bio parameter based on the vast data set collected.

The bio parameter under consideration are: Arterial Systolic and Diastolic, MAP, PA systolic, PA Diastolic, CO, Heart rate, Stroke volume, WBC, RBC, Hgb, HCT ,Iron, PLT, PH, PCO2, PO2, HCO3, SaO2 , Na, K, Cl, CO2, Bun, Cr, Gluc, HGB (A1C),TBiLi, LDL, HDL.

This study hopes to demonstrate the connection between blood color pigmentation and certain bio parameters for simplifying monitoring procedure and particular home monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18
2. Patients with cardiovascular disease and/or with diabetes mellitus type I or II and/or with COPD.
3. Patients receiving coronary artery bypass with or without valve repair.
4. Able to sign an informed consent.

Exclusion Criteria:

1. Refusal to sign an informed consent and to participate in the study.
2. Participant plans to enroll in another other clinical trial of an investigational agent while participating in this study.
3. Below the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Smart, M.D, Principal Investigator — Chairman of the Cardiovascular Medicine Department at Morritwon Memorial Hospital and Atlantic Health; Yosef Segman, PhD, Study Chair — Cnoga Medical Ltd.; Donna Hesari, BSN, Study Director — Atlantic Health System, Department of Cardiovascular Medicine
Locations (1):
- Atlantic Health - Morristown Memorial Hospital- Cardiovascular Medicine, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website. — http://www.cnoga.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: during 2009
Groups:
- Non Invasive Monitoring: Single group of hospitalized cardiovascular patients.
  Non invasive peripheral blood monitoring: non invasive monitoring
Period: Overall Study
Arm/Group | Non Invasive Monitoring
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Non Invasive Monitoring: single group of hospitalized cardiovascular patients
Arm/Group | Non Invasive Monitoring
Number analyzed (Participants) | 94
Age, Continuous [Mean (Full Range); unit: years] — 18 years and older
  years | 51.5 [18 to 85]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  number of participants | 94
  Male | 45
  Female | 49
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the TensorTip Accuracy Against Hospital Periodical Readings.
Description: To validate the parameters with similar measures obtained with standard invasive techniques in hospitalized patients.
  Methodology:
  Eligible real time color signal obtained by the TensorTip shall be recorded simultaneously during the monitoring performed.
  An algorithm shall be designed according to the blood color distribution to each parameter and a final test shall be recorded signals.
  Statistical analysis for each parameter shall perform on the entire eligible recorded signals.
  Determination of Accuracy:
  Err = √(1/N ∑N (Ref(k)-NewDevice(k)) ^2 ) (k=1)
  For each parameter a satisfactory result is considered when Err satisfies the industry requirement.
  Results viewing Each parameter comparative study shall be presented on a (X,Y) plan versus a regression line where X - represents the results measured by TensorTip and Y - the reference results.
Time Frame: one year
Measure: Number; unit: percentage of error
Arm/Group | Non Invasive Monitoring
Number analyzed (Participants) | 94
percentage of error
  pulse | 0.6
  Blood Pressure-systolic | 7.9
  Blood Pressure-diastolic | 7.5
  Spo2 | 2.33
  PO2 | 5.99
  PCO2 | 5.3
  MAP | 6.67
  Hemoglobin | 8.9
  cardiac output | 26.9
  Hematocrit | 3.8
  RBC | 4
  O2 | 1.15
  CO2 | 4.75
  Stroke volume | 26.9
  pH | 0.03
Statistical Analysis 1: Comparison: Non Invasive Monitoring; Test type: Superiority or Other; All data in the outcome measure table is presenting the percentage of error

ADVERSE EVENTS:
Arm/Group | Non Invasive Monitoring
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No